CLINICAL TRIAL: NCT07291297
Title: Metformin Hydrochloride in Combination With Standard of Care Systemic Therapy in Previously Untreated Advanced Unresectable or Metastatic Soft Tissue Sarcoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Atrium Health Levine Cancer Institute (Other); Paula Takacs Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00138078; ONC-SAR-2401 (Other: Atrium Health)
Record Dates: First submitted 2025-12-17; First posted 2025-12-18 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Sarcoma Metastatic; Sarcoma, Soft Tissue
Keywords: Advanced Unresectable or Metastatic Soft Tissue Sarcoma; Metformin Hydrochloride
MeSH Terms: conditions — Sarcoma | interventions — Metformin

STUDY DESIGN:
Intervention Model Description: Single Arm, Metformin
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Metformin Hydrochloride ER (Other): 1000mg early release (ER) of metformin by mouth daily for 14 days, in combination with physician directed SOC systemic therapy for advanced unresectable or metastatic STS. Toleration of the starting dose of metformin at 1000mg ER daily will be assessed during an office visit with the treating provider prior to Course1-D15.
  If toleration has been deemed acceptable, the metformin dose will be increased from 1000mg ER daily to 1000mg ER twice a day starting on Course1-D15. If the participant does not meet all criteria for dose escalation, the participant will continue to receive 1000mg ER daily.
  Interventions: Drug: Metformin Hydrochloride ER

INTERVENTIONS:
Drug: Metformin Hydrochloride ER — Participants will initially take 1000mg ER of metformin by mouth daily for 14 days, in combination with physician directed SOC systemic therapy for advanced unresectable or metastatic STS.

SUMMARY:
The purpose of this research study is to see how metformin, when used in combination with standard of care (SOC) treatment for metastatic (cancer that has spread) soft tissue sarcoma can improve patient outcomes.

DETAILED DESCRIPTION:
This is a single arm, phase II, open-label study of metformin in combination with physician directed SOC first-line systemic therapy in participants with advanced unresectable or metastatic STS. Participants will continue study treatment for 5 years or until early treatment discontinuation. Metformin treatment intervention should begin no later than 4 weeks from the initiation of front-line SOC therapy.

Participants will initially take 1000mg ER of metformin by mouth daily for 14 days, in combination with physician directed SOC systemic therapy for advanced unresectable or metastatic STS. Toleration of the starting dose of metformin at 1000mg ER daily will be assessed during an office visit with the treating provider prior to Course1-D15.

Toleration of the 1000mg ER daily dose will be defined by the participant meeting all criteria below at the Course 1-Day15 (+ 7 days) study visit:

* No grade 3/4 metformin-related toxicities since initiation of metformin
* No metformin-related GI upset since initiation of metformin including diarrhea
* Acceptable organ function
* The treating provider must agree the participant has sufficiently tolerated the starting dose of the treatment intervention.

If toleration has been deemed acceptable, by meeting all criteria above as outlined, the metformin dose will be increased from 1000mg ER daily to 1000mg ER twice a day starting on Course1-D15. If the participant does not meet all criteria above for dose escalation, the participant will continue to receive 1000mg ER daily.

ELIGIBILITY:
Inclusion Criteria:

1. Advanced unresectable or metastatic/intermediate/high grade soft tissue sarcoma
2. Age ≥ 18 years at the time of enrollment
3. Initiating first line systemic therapy for advanced/metastatic disease (treatment naïve for advanced/metastatic disease)

   1. Participants who have not yet initiated first line systemic therapy: expected to initiate front-line therapy within 4 weeks of initiating metformin
   2. Participants who have previously initiated first line systemic therapy: No more than 4 weeks from initiation of first line systemic therapy
4. Adequate performance status (PS) defined as ECOG PS = 0-2
5. Adequate renal function
6. Adequate liver function
7. Individuals of childbearing potential (ICBP) must have a negative serum pregnancy test within 7 days prior to enrollment. NOTE: Individuals who may become pregnant are considered to have childbearing potential unless they are surgically sterile (have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or are postmenopausal (at least 12 consecutive months with no menses without an alternative medical cause). Metformin is known to be excreted in breast milk and should not be used by nursing mothers.
8. ICBP and partners of ICBP must not be expecting to conceive and be willing to use a highly effective contraceptive method (i.e., achieves a failure rate of <1% per year when used consistently and correctly) from the time of informed consent until 30 days after study treatment discontinuation.
9. Individuals who are having sexual relationships in which their partners may become pregnant must be willing to use condoms from the time of informed consent until 30 days after study treatment discontinuation. For a non-pregnant ICBP partner, contraception recommendations should also be considered.
10. Ability to ingest oral medications

Exclusion Criteria:

1. Already prescribed and taking metformin at time of diagnosis of advanced unresectable or metastatic disease
2. Planned enrollment on a treatment clinical trial for first line therapy
3. Breastfeeding within the duration of anticipated study treatment. NOTE: breast milk cannot be stored for future use while the mother is being treated on study.
4. History of acute or chronic metabolic acidosis including diabetic ketoacidosis, with or without coma.
5. Participants previously diagnosed with an additional malignancy must be disease-free for at least five years prior to enrollment. Exceptions include ductal carcinoma in situ (DCIS), basal cell or squamous cell skin cancer and in situ cervical or bladder cancer.
6. Treatment with any investigational drug within 14 days prior to day 1 of treatment
7. History of allergic reactions attributed to compounds of similar chemical or biologic composition to metformin. Participants receiving any medications or substances that are inhibitors or inducers of CYP450 enzyme(s) are ineligible. Lists including medications and substances known or with the potential to interact with the specified CYP450 enzyme(s) isoenzymes. Please refer to https://drug-interactions.medicine.iu.edu/MainTable.aspx for the most current information.
8. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure requiring pharmacologic treatment, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements as determined by the investigator.
9. Patients with known brain or active central nervous system (CNS) metastases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-10 (Estimated); Study Completion 2033-10 (Estimated)

PRIMARY OUTCOMES:
Number of participants surviving at 12 months | From date of metformin start to date of death, or censored at 12 months, whichever occurred first.
  12-month overall survival (OS) will be determined for each participant as a binary variable indicating whether the participant was surviving at 12 months after study enrollment. Failure occurs if the participant dies from any cause within 12 months of study enrollment (initiation of metformin).

SECONDARY OUTCOMES:
Overall survival (OS) | From date of metformin start to date of death, or censored as described; assessed for approximately 5 years.
  OS is defined as the duration of time from initiation of metformin to date of death from any cause. Surviving participants will be censored at the last known date they were alive.
Cancer specific survival | From date of metformin start to date of death, or censored as described; assessed for approximately 5 years.
  Cancer specific survival is defined as the duration of time from initiation of metformin to date of sarcoma-related death. For participants who die from causes unrelated to sarcoma, cancer-specific survival will be calculated at the date of death, with non-cancer specific death as a competing risk event. Surviving participants will be censored at the last known date they were alive.

OTHER OUTCOMES:
Metformin administration | From start of metformin treatment until last dose of study treatment; approximately 5 years
  Descriptive summary of daratumumab administration, including number of courses received and number of doses received.
Number of participants with at least one adverse event attributable to metformin | From start of metformin treatment until 30 days after last dose of study treatment; approximately 5 years
  A binary variable will be determined for each participant indicating whether the participant had at least one metformin-attributed adverse event. Adverse events will be categorized per NCI Common Terminology for Adverse Events version 5.0. Metformin attribution will be determined per treating investigator.
Number of participants with at least one serious adverse event | From start of metformin treatment until 30 days after last dose of study treatment; approximately 5 years
  A binary variable will be determined for each participant indicating whether the participant had at least one adverse event that was categorized as serious, regardless of causality. Serious is defined per the study protocol and includes events that the investigator deems serious and results in the following outcomes: death, life-threatening situation, persistent or significant disability/incapacity, requires or prolongs hospitalization, congenital anomaly/birth defect in the offspring of a study participant, suspected transmission of any infectious agent via medial product, or based upon medical judgement, may jeopardize the subject and may require medical or surgical intervention to prevent one of the afore listed outcomes from occurring.
Number of participants who discontinued study treatment due to adverse events | From start of metformin treatment until 30 days after last dose of study treatment; assessed for approximately 5 years.
  A binary variable will be determined for each participant indicating whether the participant discontinued metformin due to adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Megan Jagosky, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (2):
- United States (2):
  - Levine Cancer Institute, Charlotte, North Carolina
  - Atrium Health Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina